CLINICAL TRIAL: NCT03099239
Title: A Phase I Study of hCT-MSC, An Umbilical Cord-Derived Mesenchymal Stromal Cell Product, in Children With Autism Spectrum Disorder
Brief Title: hCT-MSCs for Children With Autism Spectrum Disorder (ASD)
Acronym: hCT-MSCs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Joanne Kurtzberg, MD (Other)
Collaborators: The Marcus Foundation (Other)
Responsible Party: Sponsor-Investigator, Joanne Kurtzberg, MD, Chief Scientific Officer, Robertson Clinical and Translational Cell Therapy Program; Director, Pediatric Blood and Marrow Transplant Program, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Pro00079421
Record Dates: First submitted 2017-03-24; First posted 2017-04-04 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Autism; Autism Spectrum Disorder; ASD
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Single hCT-MSC infusion (Experimental): Subjects 1-3 will receive a single infusion of hCT-MSCs.
  Interventions: Biological: hCT-MSC infusion
- Two hCT-MSC infusions (Experimental): Subjects 4-6 will receive two infusions of hCT-MSCs.
  Interventions: Biological: hCT-MSC infusion
- Three hCT-MSC infusions (Experimental): Subjects 6-12 will receive three infusions of hCT-MSCs.
  Interventions: Biological: hCT-MSC infusion

INTERVENTIONS:
Biological: hCT-MSC infusion — hCT-MSCs are a product of allogeneic cells manufactured from digested umbilical cord tissue that is expanded in culture, cryopreserved and banked.

SUMMARY:
The purpose of this Phase 1 study is to determine the safety of one, two, and three intravenous infusions of human umbilical cord tissue-derived mesenchymal stromal cells (hCT-MSC), administered every two months, in children with autism spectrum disorder (ASD).

DETAILED DESCRIPTION:
This study is a phase I, prospective, open-label trial designed to assess the safety of one, two, and three intravenous doses of hCT-MSC in young children with ASD. Children ages two to 11 years with ASD will be eligible to participate. All participants will receive intravenous infusion(s) of CTCs. The first cohort of three patients will receive a single dose. If there are no safety concerns, the second cohort of three patients will receive two doses, given two months apart. The third cohort will consist of six patients, each of whom will receive three hCT-MSC infusions with a two-month interval between doses. All participants will have an initial clinical evaluation to verify the diagnosis of ASD and confirm protocol eligibility. The main endpoint is safety, for which acute infusion reactions and incidence of infections will be assessed. ASD-specific outcome measures, described below, will be assessed at baseline and six months from baseline and results will be described.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 2 years to ≤ 12 years (11 years, 364 days) at the time of consent
2. Confirmed clinical DSM-5 diagnosis of Autism Spectrum Disorder using the DSM-5 Checklist with a moderate severity level of ASD as reflected by SRS score ≥ 66 and CGI-S severity score of ≥ 4.
3. Fragile X testing performed and negative; CMA and/or whole exome sequencing performed and results not linked to autism diagnosis
4. Stable on current psychiatric medication regimen (dose and dosing schedule) for at least 2 months prior to infusion of study product
5. Normal absolute lymphocyte count (≥1500/uL)
6. Participant and parent/guardian are English speaking
7. Able to travel to Duke University up to four times (baseline, every two months for subsequent infusions, and 6 months after initial infusion), and parent/guardian is able to participate in interim surveys and interviews
8. Parental consent

Exclusion Criteria:

1. General:

   1. Review of medical records indicates ASD diagnosis not likely
   2. Known diagnosis of any of the following coexisting psychiatric conditions: depression, bipolar disorder, schizophrenia, obsessive compulsive disorder associated with bipolar disorder, Tourette syndrome
   3. Screening data suggests that participant would not be able to comply with the requirements of the study procedures as assessed by the study team
   4. Family is unwilling or unable to commit to participation in all study-related assessments, including protocol follow up
   5. Sibling is enrolled in this (Duke hCT-MSC) study
2. Genetic:

   1. Records indicate that child has a known genetic syndrome such as (but not limited to) Fragile X syndrome, neurofibromatosis, Rett syndrome, tuberous sclerosis, PTEN mutation, cystic fibrosis, muscular dystrophy or a genetic defect definitively known to be associated with ASD
   2. Evaluation by geneticist (performed locally as standard of care or remotely by the study geneticist via review of available data - minimally medical records, photos, Fragile X and CMA testing) indicates a genetic cause for ASD.
3. Infectious:

   1. Known active CNS infection
   2. Evidence of uncontrolled infection based on records or clinical assessment
   3. Known HIV positivity
4. Medical:

   1. Known metabolic disorder
   2. Known abnormal thyroid function (patients with treated hypothyroidism with a normal TSH may be included)
   3. Known mitochondrial dysfunction
   4. History of unstable epilepsy or uncontrolled seizure disorder, infantile spasms, Lennox Gastaut syndrome, Dravet syndrome, or other similar chronic seizure disorder
   5. Active malignancy or prior malignancy that was treated with chemotherapy
   6. History of a primary immunodeficiency disorder
   7. History of autoimmune cytopenias (i.e., ITP, AIHA)
   8. Coexisting medical condition that would place the child at increased risk for complications of study procedures
   9. Concurrent genetic or acquired disease or comorbidity(ies) that could require a future stem cell transplant
   10. Significant sensory (e.g., blindness, deafness, uncorrected hearing impairment) or motor (e.g., cerebral palsy) impairment
   11. Impaired renal or liver function as determined by serum creatinine >1.5mg/dL or total bilirubin >1.3mg/dL, except in patients with known Gilbert's disease
   12. Significant hematologic abnormalities defined as: Hemoglobin <10.0 g/dL, WBC < 3,000 cells/mL, ALC <1000/uL, Platelets <150 x 10e9/uL
   13. Evidence of clinically relevant physical dysmorphology indicative of a genetic syndrome as assessed by the PIs or other investigators, including a medical geneticist and psychiatrists trained in identifying dysmorphic features associated with neurodevelopmental conditions.
5. Current/Prior Therapy:

   a. History of prior cell therapy b. Current or prior use of IVIG or other anti-inflammatory medications with the exception of NSAIDs c. Current or prior immunosuppressive therapy i. No systemic steroid therapy that has lasted >2 weeks, and no systemic steroids within 3 months prior to enrollment. Topical and inhaled steroids are permitted.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-06-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Infusion reactions | Assessed for a significant change at the time of each infusion, 24 hours after each infusion, 7-10 days after each infusion, 6 and 12 months after the final infusion.
  Patients will be assessed for infusion reactions.
Incidence of Infections | Assessed for a significant change at the time of each infusion, 24 hours after each infusion, 7-10 days after each infusion, 6 and 12 months after the final infusion.
  Patients will be assessed for infections.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Kurtzberg, MD, Principal Investigator — Duke University; Geraldine Dawson, PhD, Principal Investigator — Duke University; Jessica Sun, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No